CLINICAL TRIAL: NCT01914289
Title: Comparison of Resection and Radiotherapy in the Prognosis of Intrahepatic Cholangiocarcinoma Patients
Brief Title: Prognosis of Resection and Radiotherapy in the Treatment of Intrahepatic Cholangiocarcinoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, director of department of special treatment, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2013-002-02
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Prognosis; Resection; Radiotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resection (Experimental): To observe prognosis of resection of icc
  Interventions: Procedure: Resection; Radiation: Radiotherapy
- Radiotherapy (Active Comparator): To observe the prognosis of radiotherapy treatment of icc
  Interventions: Procedure: Resection; Radiation: Radiotherapy

INTERVENTIONS:
Procedure: Resection
Radiation: Radiotherapy

SUMMARY:
The purpose of this study is to confirm that prognosis of Intrahepatic Cholangiocarcinoma (ICC) with resection and radiotherapy ,to find which is safe and effective treatment.

DETAILED DESCRIPTION:
Intrahepatic Cholangiocarcinoma (ICC), the second most common primary liver cancer and constitutes 10% of primary liver malignancies.

Current therapies for the treatment of ICC are ineffective and the role of liver transplantation is not well defined.

This study reviews our experience with this tumor and looks for preoperative and pathologic indices that may help determine long term prognosis

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 17 years and <=60 years of age. confirmed case (patients with ICC) Tumors can be radical removed and resection volume was ≤50%. Criteria of liver function: Child A level, serum bilirubin ≤ 1.5 times the upper limit of normal value,alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.

No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal. Hbg ≥ 90g/L, WBC ≥ 3.000 cells/mm³,platelets ≥ 80.000 cells/mm³.

Karnofsky Performance Score performance over 60. Patients who can understand this trial and have signed information consent.

Exclusion Criteria:

* Patients who have undergone previous treatment by Resection or Radiotherapy. Patients with apparent cardiac, pulmonary, cerebronic and renal dysfunction, which may affect the treatment of liver cancer.

Patients with other diseases which may affect the treatment mentioned here. Patients with medical history of other malignant tumors. Subjects participating in other clinical trials. Extrahepatic metastasis, portal vein or other major vascular involvement. liver function: Child B C.

Patients would not sign the consent to the trial.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
the overall survival rate of each group | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Aijun, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China